CLINICAL TRIAL: NCT03451656
Title: Prospective System Analysis of Seasonal Influenza - Virus Transmission and Evolution in Basle Town
Brief Title: Prospective System Analysis of the Seasonal Influenza Virus Transmissions and Evolution in the City of Basel Basel
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-01735; me15Egli2
Record Dates: First submitted 2018-02-23; First posted 2018-03-02 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum and DNA, nasopharyngeal swamps
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The project aims to use epidemiological tools to understand the transmission and evolution of influenza viruses at an individual and population level within a small-scale city (Basel) through a combination of experimental, clinical, and mathematical advances. Investigators aim to quantitatively characterize the viral transmission using novel molecular-epidemiological tools based on whole genome sequencing.

DETAILED DESCRIPTION:
Samples will be collected such as whole blood, serum and DNA, nasopharyngeal swamps to diagnose influenza by polymerase chain reaction (PCR) and to determine colonization rates with Staphylococcus aureus and Streptococcus pneumonia. All samples except the first naso-pharyngeal swab for influenza diagnostics will be stored in a biobank and analysed in batches. Each influenza virus isolate will be sequenced using a "whole genome sequencing" approach. The viral transmission and evolution will be analysed using whole genome data for a detailed molecular and phylogenetic tree analysis, respectively. The epidemiological and geographical data will be incorporated into the phylogenetic model.

ELIGIBILITY:
Inclusion Criteria:

* Each pediatric or adult patient, which fulfill the World Health Organization (WHO) definition of Influenza like illness.
* The case definition includes an acute respiratory infection with coughing, fever ≥38°C, and start of symptoms within the last 10 days.
* Presentation of the patient with influenza-like illness on the emergency ward of the University Hospital Basel or the University Children Hospital of both Basel or a collaborating private practise.

Exclusion Criteria:

- Case definition for influenza like illness is not fulfilled

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Paediatric or adult patients fulfilling the WHO-definition of an influenza-like illness and living at Basel.
Sampling Method: Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2016-12-27 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Similarity of Influenza viruses | at baseline
  Genomic sequencing of single virus of individual patients and comparison of genetic similarity of viruses. Grouping of patients with a same virus - this includes a range of single nucleotide polymorphisms of 0-150 differences inbetween the virus population.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Egli, PD MD, Principal Investigator — Clinical Microbiology; University Hospital Basel

IPD SHARING:
Plan to Share IPD: Undecided